CLINICAL TRIAL: NCT07262281
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of HY6725 Following Single and Multiple Subcutaneous Doses in Healthy Participants
Brief Title: Evaluation of the Safety, Tolerability and Pharmacokinetics of HY6725 in Healthy Adult Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Newsoara Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Newsoara HYK Biopharmaceutical (Shanghai) Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HY6725-01-01
Record Dates: First submitted 2025-11-19; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HY6725 (Experimental): It's an injection solution. SAD part for subcutaneous dosing in 7 cohorts, including 3mg, 10mg, 30mg, 90mg, 150mg, 300mg and 450mg with only one administration on Day 1 of each cohort. MAD part for subcutaneous dosing in 3 cohorts, including 150mg, 300mg and 450mg with two administrations on Day 1 and Day 30 of each cohort.
  Interventions: Biological: HY6725
- placebo (Placebo Comparator): It's same injection solution just without active ingredient compared with HY6725. SAD part for subcutaneous dosing in 7 cohorts, including 3mg, 10mg, 30mg, 90mg, 150mg, 300mg and 450mg with only one administration on Day 1 of each cohort. MAD part for subcutaneous dosing in 3 cohorts, including 150mg, 300mg and 450mg with two administrations on Day 1 and Day 30 of each cohort.
  Interventions: Other: Placebo Control

INTERVENTIONS:
Biological: HY6725 — HY6725 is an injection solution with 120mg/ml per vial. SAD part for subcutaneous dosing in 7 cohorts, including 3mg, 10mg, 30mg, 90mg, 150mg, 300mg and 450mg with only one administration on Day 1 of each cohort. MAD part for subcutaneous dosing in 3 cohorts, including 150mg, 300mg and 450mg with two administrations on Day 1 and Day 30 of each cohort.
  Arms: HY6725
Other: Placebo Control — A vial with 1ml injection solution contain same ingredient except HY6725 compared with HY6725 solution.
  Arms: placebo

SUMMARY:
The goal of this clinical trial is to learn the safety, tolerability and pharmacokinetics of single and multiple doses of HY6725 in healthy adult participants. The main questions it aims to answer are:

* How is the safety and tolerability following administration of single and multiple doses of HY6725 in healthy adult participants?
* What is the PK character of HY6725 following administration of single and multiple doses of HY6725 in healthy adult participants?

Researchers will compare HY6725 to a placebo (a look-alike substance that contains no drug) to see if HY6725 is safe and well tolerated.

Participants will take HY6725 or a placebo once or twice in single dose group or multiple dose group. And will be follow-up until Day 150.

DETAILED DESCRIPTION:
The rationale of the study is HY6725 is a novel, fully human monoclonal antibody engineered to simultaneously neutralize human TSLP and IL-33. Given the overlapping, synergistic, and compensatory roles of TSLP and IL-33 in the pathogenesis of asthma and COPD-as well as in other chronic type 2 inflammatory diseases-simultaneous inhibition offers a promising therapeutic strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants must be 18 to 55 years of age, inclusive, at the time of signing the informed consent.
2. Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, vital sign assessments, laboratory tests, and 12-lead ECGs.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures
4. BMI of 18 to 32 kg/m2; and a total body weight>50 kg.
5. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the informed consent and in this protocol.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary (but excluding resolved childhood asthma), gastrointestinal (but excluding resolved gall bladder and appendix removal), cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. History of HIV infection, hepatitis B, hepatitis C or syphilis; positive testing for HIV, hepatitis B, HCVAb or serological reaction of syphilis

   • For hepatitis B, all participants must undergo testing for HBsAg, HBcAb, and HBsAb.
   * Participants who are negative for all 3 serology tests may be eligible.
   * Participants who are HBsAg positive will be excluded.
   * HBsAg negative, HBcAb positive, and HBsAb negative particpants are to be excluded from the study.
   * Participants who are HBsAg negative, HBcAb negative and HBsAb positive and provide documentation of prior HBV vaccination, may be eligible for the study and will not require HBV DNA monitoring during the study.
   * Participants who are HBsAg negative, HBcAb negative and HBsAb positive without documentation of prior HBV vaccination AND participants who are HBsAg negative, HBcAb positive, and HBsAb positive, will have HBV DNA assessed at screening.

     * If HBV DNA is detectable, participants will be excluded.
     * If HBV DNA is not detectable, participants may be eligible.
3. History of severe allergic or anaphylactic reaction to a therapeutic drug.
4. History of recent active infections within 28 days prior to the screening visit.
5. History of recent iron deficiency requiring treatment within 3 months before the first dose of study intervention.
6. Participants with a fever within 48 hours prior to dosing.
7. Participants who are QFT-G test positive will be excluded.
8. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
9. Use of prescription medications within 14 days and over-the-counter medications within 7 days before the first dose of study intervention (except for the ones listed in section 6.9.2 ) . However, there can be some investigator discretion to allow some medication. (Refer to Section 6.9 Prior and Concomitant Therapy for additional details).
10. Recent exposure to live vaccines within 28 days of the screening visit.
11. Known exposure to anti-TSLP or IL-33 or any type of anti-TSLP or anti-IL-33 therapy.
12. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
13. A positive urine drug test.
14. A positive pregnancy test.
15. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and non clinically significant results may be inclusionary at the opinion of the investigator.
16. Baseline 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (e.g. baseline QTcF interval >450 msec, complete LBBB, signs of an acute or indeterminate -age myocardial infarction, ST-T interval changes suggestive of myocardial ischemia, second or third-degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate corrected- using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF or QRS values should be used to determine the participant's eligibility. Computer interpreted- ECGs should be overread by a physician experienced in reading ECGs before excluding participants.
17. Participants with of ANY following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:

    * AST or ALT level ≥1.5 x ULN;
    * Total bilirubin level ≥1.5 x ULN; participants with a history or suspected of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.
    * And other clinically significant laboratory results in the opinion of the investigator.
18. History of drug or alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit= 240 mL beer, 30 mL of 40% spirit, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine). And participants with >2 cigarettes per day intake and with >5 cigarettes per week intake.
19. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 30 days prior to dosing.
20. History of sensitivity to heparin or heparin-induced thrombocytopenia.
21. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
22. Investigator site staff or the sponsor employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Safety data including incidence and severity of TEAEs, SAEs, change from baseline in vital signs, lab values and ECG parameters. | From signing informed consent form to the end of study at Day 150.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | From Day1 predose to Day 150.
Area under the plasma concentration versus time curve (AUC) | From Day1 predose to Day 150.
Time to maximum concentration (Tmax) | From Day1 predose to Day 150.
Plasma half-life time (T1/2) | From Day1 predose to Day 150.

CONTACTS AND LOCATIONS:
Overall Officials: Weifen Zhou, Dr., Study Director — Newsoara Biopharma Co., Ltd.
Locations (1):
- Nucleus Network Pty Ltd., Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No